CLINICAL TRIAL: NCT05090371
Title: A Randomized, Open Label, Multi-center, Active-comparator Study to Assess Efficacy, Safety & Tolerability of Ofatumumab 20mg sc Monthly Versus Continued Current Therapy in Relapsing-remitting Multiple Sclerosis After Elevation of Serum Neurofilament Light Levels (SOSTOS)
Brief Title: A Multicenter Study of Continued Current Therapy vs Transition to Ofatumumab After Neurofilament (NfL) Elevation
Acronym: SOSTOS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMB157GUS09
Record Dates: First submitted 2021-10-12; First posted 2021-10-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Ofatumumab; Multiple Sclerosis; Relapsing-Remitting Multiple Sclerosis; adult; OMB157; RRMS; MS; secondary progressive MS; relapse
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Recurrence | interventions — ofatumumab

STUDY DESIGN:
Intervention Model Description: A randomized, open label, multi-center, active-comparator study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ofatumumab (Experimental): 20 mg
  Interventions: Drug: Ofatumumab
- DMT continued therapy (Active Comparator): Participants randomized to the continued therapy arm will continue to take their disease modifying treatment (DMT) as prescribed commercially by their physician.
  Interventions: Drug: Disease modifying treatment (DMT)

INTERVENTIONS:
Drug: Ofatumumab — 3 loading doses followed by administration every 4 weeks as per label
  Arms: Ofatumumab
Drug: Disease modifying treatment (DMT) — Other DMT with approved label use for treatment which participants were on at least 6 months prior to Screening
  Arms: DMT continued therapy

SUMMARY:
This study will evaluate if relapsing-remitting MS patients that have not had a relapse in the past year would benefit from a switch to ofatumumab versus staying on their continued current therapy. This study will also look at whether an elevated serum neurofilament light (NfL) level predicts enhanced benefit from a switch to ofatumumab.

DETAILED DESCRIPTION:
This is a multicenter, prospective study of up to 150 relapsing-remitting MS participants/ The study is looking to see if patients who have not had a relapse in the past year would benefit from switching to ofatumumab.

After giving consent, participants will have a 1 week screening/qualification period. If they qualify to continue, they will start a a six month run-in period during which lab samples will be collected. Patients that are relapse-free during the run-in period will continue into next period of the study in which they will be randomized to either ofatumumab or continued therapy for the next 15 months. Every 3 out of 5 randomized participants will be selected to wear a digital study watch to collect physical activity, sleep, and vitals during this 15 month period. The study watch will be worn 24 hours a day, 7 days a week but can be removed during showers/bathing. At the end of the 15 month period, a study completion visit will be held.

The total study duration is 21 months plus 1 week for screening/qualification.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Age 18-45 years
* Diagnosis of RRMS per McDonald Criteria (2017)
* EDSS 0-5.5 (Inclusive)
* Able to obtain MRI and attend study visits at sites
* Willing to use wearable device as specified in the protocol
* Able to provide blood sample
* On a current DMT with approved label use for treatment of RRMS at least 6 months prior to Screening
* No relapse reported within 6 months prior to Screening
* Patients may enroll in the trial if they have subclinical disease activity as measured by MRI prior to enrollment. An absence of MRI activity is not exclusionary.

Exclusion Criteria:

* Primary progressive or secondary progressive phenotype
* Diseases other than multiple sclerosis responsible for the clinical or MRI presentation
* Use of experimental or investigational drugs for MS within 2 years from Screening
* Known sensitivity to gadolinium
* Central Nervous System (CNS) anomalies that are better accounted for by another disease process
* Known active malignancies
* Active chronic disease (or stable but treated with immune therapy) of the immune system other than MS
* Active infections including systemic bacterial, viral (including COVID-19) or fungal infections, known to have AIDS or tested positive for HIV antibodies
* Neurological findings consistent with Progressive Multifocal Leukoencephalopathy (PML), or confirmed PML
* IgG or IgM levels below lower limit of normal (LLN) at Screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving NEDA-3 (No Evidence of Disease Activity-3) | Months 3 to 15
  A participant is considered as achieved NEDA-3 if the participant has not had a clinical relapse (recurrence of a disease activity after a recovery), has not had an increase in disability and has no new radiological MRI activity (no new occurrences of contrast-enhancing lesions) during study Months 3 to 15.

SECONDARY OUTCOMES:
Percentage of participants with a single baseline NfL≥10pg/ml and NfL<10pg/ml achieving NEDA-3 (No Evidence of Disease Activity-3) | Months 3 to15
  Participants with a single baseline NfL≥10 pg/ml and NfL<10pg/ml will be considered as achieved NEDA-3 if the participant has not had a clinical relapse (recurrence of a disease activity after a recovery), has not had an increase in disability and has no new radiological MRI activity (no new occurrences of contrast-enhancing lesions)
Annualized relapse rate in Months 3 to 15 | Months 3 to 15
  Relapses are recurrences of a disease activity after a recovery. A confirmed MS relapse is one accompanied by a clinically relevant change in the EDSS performed by the EDSS Rater, i.e. an increase of at least 0.5 points on the EDSS score, or an increase of 1 point on two functional scores (FSs) or 2 points on one FS, excluding changes involving bowel/bladder or cerebral FS compared to the previous available rating (the last EDSS rating that did not occur during a relapse). Confirmation of MS relapse based on these definitions will be done centrally.
Percentage of participants without a worsening of their disability | Months 3 to 15
  No increase or worsening of disability
Percentage of participants with NEDA (No Evidence of Disease Activity) - Clinical | Months 3 to 15
  A participant is considered as achieved NEDA-clinical is no clinical relapse or disease progression (by EDSS) has occurred.
Percentage of participants with NEDA (No Evidence of Disease Activity) - Radiological | Months 3 to 15
  A participant is considered as achieved NEDA-radiological if the participant has has no new radiological MRI activity (no new occurrences of contrast-enhancing lesions) during study Months 3 to 15.
Mean change in The Symbol-Digit Modality Test | Baseline, Months 3 and 15
  This test measures cognition in patients with MS. Patients are asked to substitute a number, either orally or written, for randomized presentations of geometric figures.
Mean change in the Time 25 Foot Walk | Baseline, Months 3 and 15
  This is a test of mobility and leg function. The patient is instructed to one end of a marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time to complete the test is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is performed again when the patient is directed to walk back the same distance. A walking device is permitted during this test.
Mean change in the 9 Hole Peg Test | Baseline, Months 3 and 15
  This is a test of upper extremity function. The patient is seated at a table with a small, shallow container holding nine pegs and a wood or plastic block containing nine empty holes. The patient picks up the nine pegs one at a time as quickly as possible, puts them in nine holes and once they are in the holes, the patient removes them again as quickly as possible one at a time, replacing them into the shallow container. The total time to complete the task is recorded. This test is performed with both the dominant and non-dominant hand.
Mean change in Gd+ lesion count | Baseline, Months 3 and 15
  Increase in the number of contrast-enhancing lesions on MRI
Mean change in Gd+ lesion volume | Baseline, Months 3 and 15
  Increase in size of contrast-enhancing lesions on MRI
Mean change in T2 lesion count | Baseline, Months 3 and 15
  Increase in new T2 lesions on MRI
Mean change in T2 lesion volume | Baseline, Months 3 and 15
  Increase in size of T2 lesions on MRI
Mean change from Baseline in T1 | Baseline up to Month 15
  Presence of new or enlarged T1 lesions
Mean change in MSQOL-54 | Month 3 to Month 15
  The MSQOL-54 is health-related quality of life questionnaire that assesses the physical, mental, and social effects experienced by MS patients, as well as functional disability. It is made up for 54 questions with a total score ranging from.0 to 100. Higher scores indicate better quality of life.
Mean whole brain and regional volume loss from Baseline | Baseline up to Month 15
  Brain volume loss is a marker of progressive loss of brain structure and function. It is a predictor of disability progression.
Percentage of participants reporting treatment emergent adverse events (TEAEs) and serious adverse events | Baseline up to Month 15
  Adverse events (TEAEs) and serious adverse events will be reported at each visit

CONTACTS AND LOCATIONS:
Locations (43):
- United States (37):
  - Alabama Neurology Associates PC, Birmingham, Alabama
  - North Central Neurology Associates PC, Cullman, Alabama
  - Radiant Research Chandler, Chandler, Arizona
  - Arizona Neuroscience Research LLC, Phoenix, Arizona
  - University of California at Los Angeles, Torrance, California
  - Neurology of Central FL Res Ctr, Altamonte Springs, Florida
  - S And D Clinical Research, Cape Coral, Florida
  - Homestead Assoc In Research Inc, Homestead, Florida
  - Neurology Associates PA, Maitland, Florida
  - Orlando Health Clinical Trials, Orlando, Florida
  - Emerald Coast Neurology, Pensacola, Florida
  - University Of South Florida, Tampa, Florida
  - Kootenai Health, Coeur d'Alene, Idaho
  - Neuro Medial Clinic of Central Louisiana, Alexandria, Louisiana
  - International Neurorehab Institute, Lutherville, Maryland
  - Reliant Medical Group, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Memorial Healthcare, Owosso, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St Barnabas Medical Center, Livingston, New Jersey
  - Jersey Shore University Medical Ctr, Neptune City, New Jersey
  - SUNY Upstate Medical Center, Syracuse, New York
  - University Of NC At Chapel Hill, Chapel Hill, North Carolina
  - Piedmont HealthCare, Charlotte, North Carolina
  - Velocity Clinical Research, Raleigh, North Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Sibyl Wray MD Neurology PC, Knoxville, Tennessee
  - Clinical Trial Network, Houston, Texas
  - Neuro Mind Clinical Trials Ltd Co, Katy, Texas
  - Covenant Medical Group, Lubbock, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Tranquil Clinical Research, Webster, Texas
  - Sentara Neuroscience Institute, Virginia Beach, Virginia
  - Evergreen Health Multiple Sclerosis Center, Kirkland, Washington
  - Swedish Medical Center, Seattle, Washington
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (6):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Burnaby, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Granby, Quebec
  - Novartis Investigative Site, Lévis, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com